CLINICAL TRIAL: NCT05554692
Title: Peripheral and Central Contributions to Auditory Temporal Processing Deficits and Speech Understanding in Older Cochlear Implantees
Brief Title: Peripheral and Central Influences on Auditory Temporal Processing & Speech Perception in Older Cochlear Implantees
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Matthew Goupell, Professor, Department of Hearing and Speech Sciences, University of Maryland, College Park
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1781406; R01DC020316 (NIH)
Record Dates: First submitted 2022-08-31; First posted 2022-09-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss; Cochlear Hearing Loss; Hearing Loss, Sensorineural; Aging
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Enrolled Participants - Older adults with cochlear implants (Experimental): Individuals who already use at least one cochlear implant.
  Interventions: Diagnostic Test: Diagnostic tests of cochlear implant function
- Enrolled Participants - Adults with typical hearing (Other): Control group to provide baseline or comparison data
  Interventions: Diagnostic Test: Diagnostic tests of auditory function

INTERVENTIONS:
Diagnostic Test: Diagnostic tests of cochlear implant function — Because the subjects in the study will use CI devices that they have already received as part of their standard-of-care treatment, the medical device itself is not an intervention for the purposes of this study. The intervention here will be to carry out diagnostic tests of CI function. This will include perceptual tests of temporal discrimination and speech understanding.
  Arms: Enrolled Participants - Older adults with cochlear implants
Diagnostic Test: Diagnostic tests of auditory function — The intervention here will be to carry out diagnostic tests of hearing. This will include perceptual tests of temporal discrimination and speech understanding.
  Arms: Enrolled Participants - Adults with typical hearing

SUMMARY:
Older adults who use cochlear implants to address hearing loss show wide variation in benefit. This research investigates the role of normal aging, the health of peripheral and central auditory pathways, and positioning of the cochlear implant electrode array in contributing to this variability. A range of input types from simple auditory signals to spoken sentences is used to examine these questions.

DETAILED DESCRIPTION:
This research aims to understand age-related temporal processing in older cochlear-implant (CI) users. The overall objective is to disentangle the peripheral and central contributions to age-related temporal processing deficits in this population. The central hypothesis is that age-related speech perception deficits are explained by unique contributions from peripheral and central auditory functions, significantly affecting outcomes in older CI users.

The central hypothesis will be tested by determining (1) the extent to which temporal processing of simple signals from single-electrode stimulation can be explained by aging and the peripheral electrode-to-neural interface; (2) the extent to which speech perception can be explained by aging and the peripheral electrode-to-neural interface; (3) the extent and manner in which central auditory compensation overcomes peripheral processing deficits that contribute to age-related performance declines in CI subjects.

Outcome measures collected in this project include behavioral measures of speech and auditory perception and electrophysiological responses.

Also collected are questionnaire-based reports of history of CI device use, cognitive screening measures, and imaging-based information regarding electrode placement in the cochlea.

Better understanding of the locus of age-related temporal processing deficits in this population will aid in developing age-specific guidance regarding CI candidacy, programming, and rehabilitation, thereby improving expected benefit and quality of life.

ELIGIBILITY:
For Cochlear Implant arm:

Inclusion Criteria:

* cochlear implant in one or both ears
* post-lingual onset of deafness
* 1+ years cochlear implant experience
* use of Cochlear-brand implants
* implanted after 2004

Exclusion Criteria:

* use of non-Cochlear-brand cochlear implants
* no use of oral language
* pregnant women are not eligible for the imaging portion of the study.
* residual acoustic hearing with unaided thresholds <90 dB HL at more than two standard audiometric frequencies
* other known disability or neurological disorder

For Typical Hearing arm:

Inclusion Criteria:

* audiometrically normal hearing, near-normal hearing, or mild/moderate hearing loss.

Exclusion Criteria:

* severe hearing loss
* history of neurological disorders
* history of middle-ear disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Perceptual forward-masking recovery | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Basic measurement of temporal processing - A masker stimulus encountered before a probe/target stimulus can affect the perception of the probe stimulus to a greater/lesser degree depending on their separation in time and their absolute and relative levels. Percent correct discrimination as a function of time separation and level manipulations, as measured from a behavioral response, will be reported.
Perceptual gap detection thresholds | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Basic behavioral measurement of temporal processing - The ability to detect a silent gap within a stimulus typically varies depending on frequency and level characteristics of the stimulus in which the gap is embedded and also with the hearing history and age of the listener. Gap detection threshold is the shortest gap duration that can be reliably detected under a given set of conditions and is typically reported in milliseconds.
Perceptual duration discrimination thresholds | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Basic measurement of temporal processing - Perceptual duration discrimination thresholds summarize a listener's ability to tell apart stimuli that differ in temporal extent. Percent correct discrimination as a function of duration difference, overall stimulus duration, and level manipulations, as measured from a behavioral response, will be reported.
Perceptual amplitude discrimination thresholds | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Basic measurement of auditory processing - Perceptual amplitude discrimination thresholds summarize a listener's ability to tell apart stimuli that differ in level. Percent correct discrimination as a function of level difference size and average level, as measured from a behavioral response, will be reported.
Speech perception | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Word discrimination, consonant, vowel, and sentence perception tests. The ability to discriminate between and identify recorded words, phonemic contrasts, and sentences will be assessed behaviorally. Results are reported in terms of percent correct words or phonemes.
Amplitude modulation detection performance | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Measure of ability to perceive amplitude modulation using modulation depth thresholds. Amplitude modulation detection performance summarizes a listener's ability to detect the presence of slower-changing amplitude variations applied to a faster-varying carrier signal. The modulation depth of the resulting combined signal can vary between 0 to 100% of the carrier signal with larger values indicating more extreme amplitude fluctuation. This research reports on the amount of modulation that can be detected as a function of different modulator and carrier frequencies, as well as overall stimulus level, as assessed via behavioral report.

SECONDARY OUTCOMES:
Electrically evoked compound action potential (ECAP) | Time Frame: Post-treatment - after at least 1 year use of a cochlear implant if CI user. Not collected from NH listeners. This measure will be collected once within a 6-month time period for each participant.
  ECAP amplitude growth function slopes will be used to predict perceptual performance. This measure uses clinically-available software to track the growth in auditory nerve response (peak-to-peak amplitude) as input level is varied from threshold to the maximal level at which the signal is comfortably loud. The slope of input-output function will be measured for each electrode along the electrode array of each CI study participant. Steeper slopes (measured in microvolts/current unit) will be interpreted as indicating better neural health of the associated auditory neurons.
Electrically evoked compound action potential (ECAP) forward masking recovery | Time Frame: Post-treatment - after at least 1 year use of a cochlear implant if CI user. Not collected from NH listeners. This measure will be collected once within a 6-month time period for each participant.
  Electrophysiological measurement of auditory nerve refractory time. This measure will be used to predict perceptual performance. Detection thresholds will be measured as masker and probe inputs are varied among a fixed set of levels and the interval between masker and probe is adjusted in duration.
Electrically or acoustically evoked auditory brainstem response (ABR) - Wave V amplitude | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Wave V from the ABR is a reflection of brainstem/midbrain processing. We will measure Wave V amplitude (microV) as the masker and probe levels and masker-to-probe interval are varied. This will be used to predict perceptual performance.
Electrically or acoustically evoked auditory brainstem response (ABR) - Wave V latency | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Wave V from the ABR is a reflection of brainstem/midbrain processing. We will measure Wave V latency (ms) as the masker and probe levels and masker-to-probe interval are varied. This will be used to predict perceptual performance.
Cortical auditory evoked potential - N1 and P2 amplitude | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Cortical (N1 and P2) amplitude (microV) in response to sound will be used to predict perceptual performance. This is an obligatory response from the auditory cortex that indicates sound detection.
Cortical auditory evoked potential - N1 and P2 latency | Post-treatment - after at least 1 year use of a cochlear implant if CI user. No required time frame for NH comparison listeners. This measure will be collected once within a 6-month time period for each participant.
  Cortical (N1 and P2) latency (ms) in response to sound will be used to predict perceptual performance. This is an obligatory response from the auditory cortex that indicates sound detection. There is evidence that this latency varies as a function of aging.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Goupell, PhD, Principal Investigator — University of Maryland, College Park; Samira B. Anderson, PhD, Study Director — University of Maryland, College Park; Sandra Gordon-Salant, PhD, Study Director — University of Maryland, College Park
Locations (1):
- University of Maryland, College Park, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data that document, support, and validate research findings will be made available when the main findings have been accepted for publication. De-identified data relevant to the project will be disseminated to researchers on and off-campus by request and review of the PI.
  After publication, research products from this project will be archived at the Digital Repository at the University of Maryland(DRUM). DRUM is a long-term, open access repository managed and maintained by the University of Maryland Libraries. Researchers and the general public can download data and code files, associated metadata and documentation, and any guidelines for reuse.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication, available for at least seven years.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee

DOCUMENTS (1):
  • Informed Consent Form (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT05554692/ICF_000.pdf